CLINICAL TRIAL: NCT03259815
Title: How Often Can Optimal Post Percutaneous Coronary Intervention (PCI) Fractional Flow Reserve (FFR) Results be Achieved? - a Randomised Controlled Trial of FFR Targeted PCI (the Target FFR Study)
Brief Title: An Evaluation of a Physiology-guided PCI Optimisation Strategy
Acronym: Target-FFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS National Waiting Times Centre Board (Other)
Responsible Party: Principal Investigator, Prof. Keith G. Oldroyd, Principal Investigator, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17/CARD/10; IRAS ID 223780 (Other: Health Research Authority)
Record Dates: First submitted 2017-08-09; First posted 2017-08-24 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease; Coronary Stenosis
Keywords: FFR Targeted PCI; Post-PCI FFR; Physiology-guided PCI Optimisation
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Care Provider
Masking Description: Operator blinded pre and post PCI coronary physiology measurements will be performed in both arms of the study.
  Post-PCI FFR results <0.90 in the interventional arm will be disclosed to the operator to allow further intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIOS Intervention Group (Experimental): Operator-blinded pre and post-PCI coronary physiology measurements will be recorded. If FFR is <0.90, the result will be disclosed to the operator and a hyperaemic pressure wire pullback will be performed during a standard peripheral intravenous adenosine infusion (140mcg/kg/min).
  The operator will then follow the PIOS protocol to attempt to obtain the target optimal post-PCI FFR result.
  Interventions: Procedure: P.I.O.S.; Diagnostic Test: Pre and post-PCI coronary physiology measurements
- Control Group (Active Comparator): Operator-blinded pre and post-PCI coronary physiology measurements will be recorded and the angiographically defined result will be accepted.
  Interventions: Diagnostic Test: Pre and post-PCI coronary physiology measurements

INTERVENTIONS:
Procedure: P.I.O.S. — Physiologically-Guided Incremental Optimisation Strategy
  Arms: PIOS Intervention Group
Diagnostic Test: Pre and post-PCI coronary physiology measurements — Pre and post-PCI coronary physiology measurements will be performed but not disclosed to the operator

SUMMARY:
There has recently been renewed interest in the measurement of post percutaneous coronary intervention (PCI) Fractional Flow Reserve (FFR). Previous studies have suggested that post-PCI FFR values ≥0.90 are associated with better clinical outcomes for patients but the available data suggest that despite angiographically satisfactory results, this is actually achieved in less than 40% of cases.

The main mechanisms for sub-optimal post-PCI FFR measurements have been proposed to be suboptimal stent deployment, unmasking of a second lesion in the target vessel post PCI, residual diffuse disease in the untreated segments and pressure drift (a technical artefact of pressure wire technology).

Using post-PCI FFR to guide stent optimisation and/or further intervention in the target vessel has been shown to increase the frequency of achieving optimal post-PCI FFR results (and therefore presumably better clinical outcomes). However, there are additional costs involved in the routine use of post-PCI FFR and it is not clear just how often it is even possible to increase the initial post-PCI FFR to ≥0.90. This uncertainty means that it is currently difficult to either recommend the routine use of post-PCI FFR or justify its cost.

The investigators propose a prospective study to assess the feasibility of achieving post-PCI FFR ≥0.90 during standard PCI procedures in consecutive patients. The study would also attempt to elucidate the mechanisms for sub-optimal FFR results when they occur. The investigators anticipate using the data from this developmental study to support a subsequent funding application for a definitive phase 3 study of the impact of FFR targeted PCI on clinical outcomes.

DETAILED DESCRIPTION:
Original hypothesis

A simple Physiology-guided Incremental Optimisation Strategy (PIOS) can increase the proportion of patients undergoing PCI in whom a post-PCI FFR ≥0.90 can be achieved from 40% to 60%.

Experimental details and design of proposed investigation

Overall aim:

A randomised controlled trial of a physiology-guided optimisation strategy to determine the feasibility of increasing the proportion of post-PCI FFR measurements ≥0.90 in a consecutive series of patients undergoing standard PCI procedures.

Study Population:

260 consecutive patients with stable angina referred for invasive management to the cardiac catheterisation lab who have been selected to undergo PCI based on either angiographic appearances or prior FFR assessment. Patients will be caffeine free for >12 hours pre-procedure.

Methods/Design:

Informed consent will be obtained prior to cardiac catheterisation in all potential subjects conforming to the inclusion and exclusion criteria.

Patients will then be randomised to one of two groups (described below) and PCI will be performed, using a pressure guidewire, according to standard practice at the Golden Jubilee National Hospital (including lesion pre-dilation and post-dilation of the stented segment).

Group 1 (PIOS Group):

Operator-blinded coronary physiology measurements will be recorded pre and post PCI.

If the post-PCI FFR is ≥0.90, no further intervention will be performed and the procedure is considered complete.

If post-PCI FFR is <0.90, the result will be disclosed to the operator and a hyperaemic pressure wire pullback during a standard peripheral intravenous adenosine infusion (140mcg/kg/min) will be performed. Depending on the result the operator would then have the following options:

A. If there is a step-up of ≥0.05 across the stented segment(s) further post-dilatation with a 0.25 - 0.50mm larger non-compliant balloon to at least 18 atmospheres should be performed followed by repeat FFR. Alternatively, the operator may choose to employ intracoronary imaging (IVUS or OCT) to guide post-dilation/optimisation of the stented segment.

B. If there is a step-up of ≥0.05 across a relatively focal (<20mm) unstented segment which is technically suitable for further stenting then a further stent should be implanted followed by repeat FFR.

C. If the FFR remains <0.90 after steps A +/- B, a further FFR pullback will be performed. If the criteria for Step B are again met, one additional stent may be deployed and a final FFR pullback performed. Following this, the FFR result will be accepted.

D. If the residual pressure gradient is interpreted to reflect diffuse atherosclerosis with no focal step-ups, the result is accepted.

E. At the end of the procedure the pressure wire sensor will be withdrawn to the tip of the guiding catheter and compared with the aortic pressure. A pressure drift of ≤0.03 will be accepted and the final FFR result adjusted accordingly.

F. If there is a drift of ≥0.04, the wire should be re-equalised and the final FFR measurement be repeated.

G. The patients will have their demographics and procedure details recorded. All patients will be asked to complete follow-up questionnaires at 3 months.

Group 2 (Control Group):

Pre and post-PCI coronary physiology measurements will be recorded but not disclosed to the operator. The angiographically defined result will be accepted. The patients will have their demographics and procedure details recorded. All patients will be asked to complete follow-up questionnaires at 3 months.

Expected value of results

1. Confirmation that the proposed PIOS protocol significantly increases the proportion of patients obtaining a physiologically optimal post-PCI result will demonstrate the feasibility of this strategy and should lead to an increase in post-PCI pressure wire usage to achieve physiologically optimal results for patients.

   The investigators hypothesise that the PIOS intervention can increase the proportion of patients achieving this target from 40% to 60% and believe that an increment of at least this magnitude would be necessary to make a future larger study with both patient-oriented clinical (target vessel failure) and health care system (resource utilisation) outcomes acceptable to the interventional cardiology community and potential funders.
2. The secondary outcome measures, albeit underpowered for clinical outcomes in this study, will hopefully still give a signal that achieving a target post-PCI FFR ≥0.90 does yield objective benefits for patients. This could then form the basis for a larger phase 3 trial to confirm improved clinical outcomes and cost- effectiveness of FFR-targeted PCI

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age with coronary artery disease (including stable angina and stabilised non-ST-elevation myocardial infarction (NSTEMI)) who are able to provide informed consent.

Exclusion Criteria:

* PCI in a coronary artery bypass graft
* PCI to an in-stent restenosis (ISR) lesion
* PCI to a target artery providing Rentrop grade 2 or 3 collateral blood supply to another vessel
* Inability to receive adenosine (for example, severe reactive airway disease, marked hypotension, or advanced atrioventricular block without pacemaker).
* Recent (within 1 week prior to cardiac catheterization) ST-segment elevation myocardial infarction (STEMI) in any arterial distribution (not specifically target lesion).
* Severe cardiomyopathy (ejection fraction <30%).
* Renal insufficiency such that an additional 20 to 30 mL of contrast would, in the opinion of the operator, pose unwarranted risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a final post-PCI FFR result ≥0.90 | 1 day
  The proportion of patients with a final post-PCI FFR result ≥0.90 will be compared between the randomised groups

SECONDARY OUTCOMES:
The proportion of patients with final post-PCI FFR ≤0.80 | 1 day
  The proportion of patients with a final post-PCI FFR result ≤0.80 will be compared between the randomised groups
Change from baseline in self-reported health outcomes at 3 months using a disease-specific quality of life measurement tool. | 3 months
  Patients will complete the Seattle Angina Questionnaire (SAQ) at baseline pre-procedure and again at 3 months post PCI
Change from baseline in self-reported health outcomes at 3 months using a generic quality of life measurement tool. | 3 months
  Patients will complete the EQ-5D questionnaire at baseline pre-procedure and again at 3 months post PCI
The rate of target vessel failure (TVF) and its component features at 3 months. | 3 months
  Component features of TVF include cardiac death, myocardial infarction, stent thrombosis, unplanned rehospitalisation with target vessel revascularisation.
The rate of target vessel failure (TVF) and its component features at 1 year. | 1 year
  Component features of TVF include cardiac death, myocardial infarction, stent thrombosis, unplanned rehospitalisation with target vessel revascularisation.
Change from baseline in the FFR following PCI | 1 day
  The difference between measurements of Fractional Flow Reserve taken in the target vessel pre- and post-PCI
The proportion of patients with final post-PCI dPR ≥0.90 | 1 day
  The proportion of patients with a final post-PCI Diastolic Pressure Ratio (dPR) value ≥0.90
Change from baseline in the Diastolic Pressure Ratio (dPR) following PCI | 1 day
  The difference between measurements of the Diastolic Pressure Ratio taken in the target vessel pre and post PCI
The proportion of patients with final post-PCI RFR ≥0.90 | 1 day
  The proportion of patients with a final post-PCI Resting Full-cycle Ratio (RFR) value ≥0.90
Change from baseline in the Resting Full-Cycle Ratio (RFR) following PCI | 1 day
  The difference between measurements of the Resting Full-Cycle Ratio (the lowest Pd/Pa ratio during the whole cardiac cycle at rest) taken in the target vessel pre and post PCI
Change in TTrest following PCI | 1 day
  Change of the thermodilution-derived resting transit time (TTrest) from pre-PCI to final post-PCI value
Change in TThyp following PCI | 1 day
  Change of the thermodilution-derived hyperaemic transit time (TThyp) from pre-PCI to final post-PCI value
The proportion of patients with final post-PCI CFR value ≥2.0 | 1 day
  The proportion of patients with a final post-PCI Coronary Flow Reserve (CFR) result ≥2.0
Change from baseline in the Coronary Flow Reserve (CFR) following PCI | 1 day
  The difference between measurements of Coronary Flow Reserve taken in the target vessel pre and post PCI
The proportion of patients with final post-PCI IMR >25 | 1 day
  The proportion of patients with a final post-PCI Index of Microcirculatory Resistance (IMR) value >25
Change from baseline in the Index of Microcirculatory Resistance (IMR) following PCI | 1 day
  The difference between measurements of IMR taken in the target vessel pre and post PCI
The proportion of patients with final post-PCI IMRc >25 | 1 day
  The proportion of patients with a final post-PCI corrected Index of Microcirculatory Resistance (IMRc) value >25
Procedure Duration | 1 day
  The time required to perform the PIOS intervention procedures will be compared with those in the control group.
The cost of additional equipment employed in the experimental arm | 1 day
  The cost of additional equipment employed in the PIOS intervention (i.e. balloons/stents/intra-coronary imaging).
Fluoroscopy Dose | 1 day
  The radiation doses for the PIOS intervention procedures will be compared with those in the control group.
Contrast Material Dose | 1 day
  The contrast material doses for the PIOS intervention procedures will be compared with those in the control group.
Incidence of procedural complications such as coronary artery dissection or perforation. | 1 day
  The incidence of procedural complications such as coronary artery dissection or perforation will be recorded and compared between the two study arms

OTHER OUTCOMES:
'As Treated' analysis of the proportion of patients with a final post-PCI FFR result ≥0.90 | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the proportion of patients with final post-PCI FFR ≤0.80 | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the change from baseline in self-reported health outcomes at 3 months as assessed by the Seattle Angina Questionnaire (SAQ) | 3 months
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the change from baseline in self-reported health outcomes at 3 months as assessed by the EQ-5D questionnaire. | 3 months
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the rate of target vessel failure (TVF) and its component features at 3 months. | 3 months
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the rate of target vessel failure (TVF) and its component features at 1 year. | 1 year
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the change from baseline in the FFR following PCI | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the proportion of patients with final post-PCI dPR ≥0.90 | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the change from baseline in the dPR following PCI | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the proportion of patients with final post-PCI RFR ≥0.90 | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the change from baseline in the RFR following PCI | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the change in TTrest following PCI | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the change in TThyp following PCI | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the proportion of patients with final post-PCI CFR value ≥2.0 | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the change from baseline in the CFR following PCI | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the proportion of patients with final post-PCI IMR >25 | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the change from baseline in the IMR following PCI | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.
'As Treated' analysis of the proportion of patients with final post-PCI IMRc >25 | 1 day
  The primary efficacy analyses of the study intervention will be carried according to the 'intention to treat' principle (i.e. results will be compared between randomised groups according to the pre-specified outcome measures).
  An 'As Treated' analysis will also be performed as an additional outcome measure. This will compare patients who actually received the PIOS intervention with those who did not.

CONTACTS AND LOCATIONS:
Overall Officials: Keith G Oldroyd, MB, MD, Principal Investigator — NHS National Waiting Times Centre Board (NHS Golden Jubilee)
Locations (1):
- Golden Jubilee National Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collison D, McClure JD, Berry C, Oldroyd KG. A randomized controlled trial of a physiology-guided percutaneous coronary intervention optimization strategy: Rationale and design of the TARGET FFR study. Clin Cardiol. 2020 May;43(5):414-422. doi: 10.1002/clc.23342. Epub 2020 Feb 10. PMID 32037592
- [Result] Collison D, Didagelos M, Aetesam-Ur-Rahman M, Copt S, McDade R, McCartney P, Ford TJ, McClure J, Lindsay M, Shaukat A, Rocchiccioli P, Brogan R, Watkins S, McEntegart M, Good R, Robertson K, O'Boyle P, Davie A, Khan A, Hood S, Eteiba H, Berry C, Oldroyd KG. Post-stenting fractional flow reserve vs coronary angiography for optimization of percutaneous coronary intervention (TARGET-FFR). Eur Heart J. 2021 Dec 1;42(45):4656-4668. doi: 10.1093/eurheartj/ehab449. PMID 34279606
- [Derived] Seki R, Collison D, Ikeda K, Sonck J, Munhoz D, Bertolone DT, Ko B, Maeng M, Otake H, Koo BK, Storozhenko T, Bouisset F, Belmonte M, Leone A, Shumkova M, Ford TJ, Mahendiran T, Berry C, De Bruyne B, Oldroyd K, Sakai K, Mizukami T, Collet C. Validation of virtual fractional flow reserve pullback curves. Catheter Cardiovasc Interv. 2024 Nov;104(6):1178-1188. doi: 10.1002/ccd.31222. Epub 2024 Sep 29. PMID 39342486
- [Derived] Collison D, Copt S, Mizukami T, Collet C, McLaren R, Didagelos M, Aetesam-Ur-Rahman M, McCartney P, Ford TJ, Lindsay M, Shaukat A, Rocchiccioli P, Brogan R, Watkins S, McEntegart M, Good R, Robertson K, O'Boyle P, Davie A, Khan A, Hood S, Eteiba H, Berry C, Oldroyd KG. Angina After Percutaneous Coronary Intervention: Patient and Procedural Predictors. Circ Cardiovasc Interv. 2023 Apr;16(4):e012511. doi: 10.1161/CIRCINTERVENTIONS.122.012511. Epub 2023 Mar 28. PMID 36974680
- [Derived] Collet C, Collison D, Mizukami T, McCartney P, Sonck J, Ford T, Munhoz D, Berry C, De Bruyne B, Oldroyd K. Differential Improvement in Angina and Health-Related Quality of Life After PCI in Focal and Diffuse Coronary Artery Disease. JACC Cardiovasc Interv. 2022 Dec 26;15(24):2506-2518. doi: 10.1016/j.jcin.2022.09.048. Epub 2022 Nov 30. PMID 36543445

DOCUMENTS (2):
  • Study Protocol (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT03259815/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT03259815/SAP_001.pdf